CLINICAL TRIAL: NCT05328531
Title: The Phase Ib/II Clinical Study of the Safety, Tolerability, Pharmacokinetics and Efficacy of Genakumab for Injection in Patients With Acute Gout
Brief Title: Clinical Study of Genakumab for Injection in Patients With Acute Gout
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Collaborators: Huashan Hospital (Other); Hainan General Hospital (Other); Linyi People's Hospital (Other); The Second Affiliated Hospital of Chongqing Medical University (Other); Changhai Hospital (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Shengjing Hospital (Other); Affiliated Hospital of Nantong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Gensci048GA-Ib/II
Record Dates: First submitted 2022-03-29; First posted 2022-04-14 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Acute Gout
Keywords: acute gout
MeSH Terms: interventions — Injections

STUDY DESIGN:
Intervention Model Description: Group A : 50mg by single subcutaneous injection; Group B : 100mg by single subcutaneous injection Group C : 195mg by single subcutaneous injection;Group D : 100mg by single subcutaneous injection Group E : 195mg by single subcutaneous injection; Group F: 1ML Compound Betamethasone Injection by single intramuscular injection
Who Masked: Participant, Investigator
Masking Description: Phase II is double-blind, participants and investigators are blind.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Genakumab for injection 50mg (Ib) (Experimental): subcutaneous injection, single dose
  Interventions: Drug: Genakumab for Injection
- Genakumab for injection 100mg (Ib) (Experimental): subcutaneous injection, single dose
  Interventions: Drug: Genakumab for Injection
- Genakumab for injection 195mg (Ib) (Experimental): subcutaneous injection, single dose
  Interventions: Drug: Genakumab for Injection
- Genakumab for injection 100mg (II) (Experimental): Genakumab for injection, subcutaneous injection, single dose Placebo for Compound Betamethasone Injection, intramuscular injection, single dose
  Interventions: Drug: Genakumab for Injection
- Genakumab for injection 195mg (II) (Experimental): Genakumab for injection, subcutaneous injection, single dose Placebo for Compound Betamethasone Injection, intramuscular injection, single dose
  Interventions: Drug: Genakumab for Injection
- Compound Betamethasone Injection 1ml (II) (Active Comparator): Compound Betamethasone Injection, 1 ml, intramuscular injection, single dose Placebo for Genakumab for injection, 100mg, subcutaneous injection, single dose
  Interventions: Drug: Placebo for Genakumab for Injection

INTERVENTIONS:
Drug: Genakumab for Injection — 150 mg/1ml/bottle
  Arms: Genakumab for injection 100mg (II); Genakumab for injection 100mg (Ib); Genakumab for injection 195mg (II); Genakumab for injection 195mg (Ib); Genakumab for injection 50mg (Ib)
Drug: Placebo for Genakumab for Injection — The placebo contains other excipients except Genakumab, and its appearance is consistent with that of Genakumab for injection
  Arms: Compound Betamethasone Injection 1ml (II)

SUMMARY:
To evaluate the safety and tolerability of single subcutaneous injection of Genakumab for Injection in patients with acute gout

DETAILED DESCRIPTION:
Phase Ib: single arm, open lable, single dose, dose escalation,design. There are 3 dose groups with 10 participant s in each group.

Phase II: randomized, double-blind, active control design.There are 2 dose groups of Genakumab for Injection with 30 participant s in each group and 1 group of Compound Betamethasone Injection with 30 praticipants.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, 18 years ≤ age ≤65 years
* Meeting the American College of Rheumatology (ACR) 2015 preliminary criteria for the classification of acute arthritis of primary gout
* Contraindication, intolerance or lack of efficacy for NSAIDs and/or colchicine
* Body mass index of less than or equal to 45 kg/m2
* Onset of current acute gout flare within 5 days prior to study entry
* Baseline pain intensity ≥ 50 mm on the 0-100 mm visual analog scale (VAS)
* History of gout flare prior to study entry

Exclusion criteria:

* evidence/suspicion of infectious/septic arthritis, or other acute inflammatory arthritis
* Presence of severe renal function impairment
* Use of specified pain relief medications or biologics ( corticosteroids, narcotics, paracetamol/acetominophen, ibuprofen, colchicine, IL-blocker, and tumor necrosis factor inhibitor) within specified periods prior to study entry
* Live vaccinations within 3 months prior to randomization
* Requirement for administration of antibiotics against latent tuberculosis (TB)
* Any active or recurrent bacterial, fungal, or viral infection
* QTc>450ms for male, QTc>470ms for female

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2021-05-22 (Actual); Primary Completion 2022-06-09 (Actual); Study Completion 2022-06-09 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | baseline, 24hours, 48hours, 120hours, Day 7, Day 14, Day 21, Day 28, Day 56, Day 84, Day 112
  Blood samples will be collected at indicated time points for pharmacokinetic analysis.
pain intensity change from baseline to 72 hours post dose as measured on a 0-100 mm Visual Analog Scale (VAS) | 72 hours post-dose
  0-100 mm Visual Analog Scale(VAS): 0= no pain and 100= severe pain

SECONDARY OUTCOMES:
Percentage of Participants With Treatment Emergent Adverse Events (TEAEs) | up to 16 weeks
  Adverse events (AEs) were defined as any unfavourable and unintended diagnosis, symptom, sign (including an abnormal laboratory finding), syndrome or disease which either occurs during study, having been absent at baseline, or, if present at baseline, appears to worsen. Serious adverse events (SAEs) were defined as any untoward medical occurrences that result in death, are life threatening, require (or prolong) hospitalisation, cause persistent or significant disability/incapacity, result in congenital anomalies or birth defects, or are other conditions which in judgement of investigators represent significant hazards
High Sensitivity C-reactive Protein (hsCRP) | at 72 hours and 7 days, 4, 8 and 12 weeks post-dose
  High sensitivity C-reactive protein (hsCRP) was determined in serum at all visits (except Visit 2 and Visit 4 ) in order to identify the presence of inflammation, to determine its severity, and to monitor response to treatment.

OTHER OUTCOMES:
Immunogenicity | baseline, Day 14, Day 28, Day 56, Day 84, Day 112
  The incidence of anti-drug antibodies (ADA) and the incidence of neutralizing antibody

CONTACTS AND LOCATIONS:
Overall Officials: Hejian Zou, Principal Investigator — Huashan Hospital; Jing Zhang, Principal Investigator — Huashan Hospital of Fudan Univeisity
Locations (1):
- Shanghai Huashan Hospital affiliated to Fudan University, Shanghai, Shanghai Municipality, China